CLINICAL TRIAL: NCT02889822
Title: The Tolerability of Alprostadil Liposome for Injection in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Yipinhong Pharmaceutical CO.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SN-YQ-2010003
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alprostadil Liposomes for Injection (Experimental): 1. Single-dose tolerance test:10ug/20ug/50ug/100ug/200ug/300ug/400ug of Alprostadil Liposome for Injection,ivgtt,qd
  2. Multiple-dose tolerance test:100ug,ivgtt,qd,continuous administration for 7 days.
  Interventions: Drug: Alprostadil Liposomes for Injection

INTERVENTIONS:
Drug: Alprostadil Liposomes for Injection — 1. Single-dose tolerance test:10ug/20ug/50ug/100ug/200ug/300ug/400ug of Alprostadil Liposome for Injection,ivgtt,qd
  2. Multiple-dose tolerance test:100ug,ivgtt,qd,continuous administration for 7 days.

SUMMARY:
Conducted in Chinese healthy adult volunteers,the study aims to observe the safety and tolerability of single/multiple-dose administration of different doses of Alprostadil Liposome for Injection as well as to confirm the safety dose range.

DETAILED DESCRIPTION:
Conducted in Chinese healthy adult volunteers,the study aims to observe the safety and tolerability of single/multiple-dose administration of different doses of Alprostadil Liposome for Injection as well as to confirm the safety dose range.

1. Single dosing tolerability test in humans.There are 7 dose (10ug,20ug,50ug,100ug,200ug,300ug,400ug) groups in the single dosing tolerance test in healthy adult volunteers.The beginning dose of the study is 10ug,according to the dose escalation method,subjects who have successfully completed previous dose group and passed the safety assessment will enter the test of next dose group with the same method.
2. Multiple dosing tolerability test in humans.Choose the proper dosage for multiple dosing tolerance test based on the single-dose tolerance test result.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers are at least 20 years of age and no older than 40.
* BMI are at least 19.0kg/m2,and no more than 24.0kg/m2.(The weight is greater than or equal to 50kg.)Subjects who are overweight or underweight will not be inclusion.
* Subjects with normal heart rate( 60-100 beats per minute) as well as normal blood pressure(systolic blood pressure:90-120 mmHg;diastolic blood pressure:60-90 mmHg).
* Subjects with normal medical history,vital signs,physical examination and clinical examination (routine blood,routine urine,blood chemistry,coagulation function and ECG,X-ray,intraocular pressure and so on).
* A negative hepatitis B surface antigen,hepatitis C,HIV or syphilis test result.
* Subjects with the ability to communicate with investigators.Besides,subjects must be willing to remain at the study center as required per protocal to complete all visit assessments.
* Given their signed written informed consent to participate.

Exclusion Criteria:

* Subjects have brain dysfunction,mental development disorders or speech disorders that unable to communicate with investigators.
* Subjects with a history of psychiatric disease or drug dependence in the past 2 years.
* Subjects with a medical history about cardiac,liver,renal,digestive system or neurological.
* Subjects with the family history of diabetes,the history of pancreatitis,cholelithiasis or asthma.
* Subjects significantly abuse alcohol or tobacco.
* Drink in 24 hours before post-dosing of study drug.
* Subjects who had taken medications within 2 weeks.
* Subjects who had suffer from exsanguine or donated blood over 200ml will be excluded.
* Subjects who participate in other clinical trials within 3 months will be excluded.
* History of hypersensitivity or allergy to any of the study drugs or to drugs of similar chemical classes.
* Subjects with a history of fainting.
* Subjects who had infected for unknown reason.
* Subjects with interstitial pneumonia.
* Subjects with glaucoma or intraocular pressure with hyperthyroidism.
* Women who were in the mentrual period.
* Women who are pregnant or lactating.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety assessment of Alprostadil Liposome for Injection | 14 days
  The safety assessment for this study include:
  1. Adverse event（AEs）
  2. Change from baseline in physical examination,vital signs,laboratory examinations
  3. Local irritation symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Zeyuan Liu, Principal Investigator — The Affiliated Hospital of Academy of Military Medical Sciences
Locations (1):
- The Affiliated Hospital of Academy of Military Medical Sciences, Beijing, China